CLINICAL TRIAL: NCT06695481
Title: Comparison of Combined Versus Conventional Radiofrequency Thermocoagulation for Lumbar Facet Joint Pain Management: a Retrospective Study
Brief Title: Radiofrequency Treatments for Lumbar Facet Joint Pain Management
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tugce Yavuz, Medical Doctor, Hacettepe University
Other Study IDs: 2023/13-08
Record Dates: First submitted 2024-07-22; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain; Zygapophyseal Joint Arthritis
Keywords: Pulsed Radiofrequency Treatment; Radiofrequency Ablation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conventional: In this group, only patients who had facet joint medial branch conventional RF applied to the patients who benefited after diagnostic injection into the facet joint were selected.
  Interventions: Procedure: Conventional RF
- Combined: This group was selected retrospectively from patients who benefited from diagnostic injection into the facet joint and who underwent pulsed rf in addition to facet joint medial branch conventional rf.
  Interventions: Procedure: Combined RF

INTERVENTIONS:
Procedure: Conventional RF — The conventional RF group consists of patients who received medial branch RF with a duration of 2 minutes, at 80̊ C temperature, and 7 Volts.
  Groups: Conventional
Procedure: Combined RF — In the combined RF group, treatment was initiated first with a conventional RF duration of 2 minutes at a temperature of 80̊ C at 7 Volts. Then, pulsed RF duration was applied for 6 minutes at a temperature of 42 C at 45 Volts, with a pulse frequency of 2 Hz and a width of 20 ms.
  Groups: Combined

SUMMARY:
In this study, investigators compared the effectiveness of medial branch conventional radiofrequency application and combined radiofrequency application in patients with lumbar facet joint disease , focusing on pain scores. The combined radiofrequency application, a sequence of pulsed radiofrequency and conventional radiofrequency , has been shown to be successful in treating neck pain and headache. These findings are of significant importance in the field of pain management and spinal disorders.

DETAILED DESCRIPTION:
The treatment of chronic pain using pulsed radiofrequency (RF) has not shown any significant side effects. As a result, a combined approach of using both pulsed and conventional RF treatment in the same session has been assumed since the 2010s. This combined RF method is still widely used for pain management. The aim of this study is to compare the effectiveness of conventional RF with the combined RF method as a medial branch RF method for the management of lumbar facet joint pain.The study involved patients who had undergone medial branch denervation for lumbar facet joint pain and had medical records available. This study was conducted retrospectively by examining the study data. Patients with missing data were excluded from the study.

Patients underwent a fluoroscopy-guided selective medial branch nerve block using 2% lidocaine 0.5ml before treatment. After 30 minutes, they were asked if there was a 50% reduction in pain intensity.The conventional RF group consists of patients who received medial branch RF with a duration of 2 minutes, at 80̊ C temperature, and 7 Volts. In the combined RF group, treatment was initiated first with a conventional RF duration of 2 minutes at a temperature of 80̊ C at 7 Volts. Then, pulsed RF duration was applied for 6 minutes at a temperature of 42 C at 45 Volts, with a pulse frequency of 2 Hz and a width of 20 ms.After procedure In the outpatient clinic, experienced pain specialists recorded NRS (Numeric Rating Scale) and DN4 (Douleur Neuropathic 4 Questions) scores at the 6th and 12th-month follow-up appointments after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 40 - 90 years of age
* Patients with low back pain for more than three months and did not respond to conservative treatment

Exclusion Criteria:

* Patients who underwent facet joint medial branch RF treatment previously
* Patients had additional interventional pain treatment or lumbar surgery within one year of the procedure
* Patients had radicular and significant disc pathology, psychiatric diseases or mental problems, malignancies
* Patients of one year follow-up could not be assessed entirely in the system

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are clinically diagnosed with lumbar facet joint pain after getting a pain reduction of over 50% following a selective diagnostic block (0.5 ml 2% lidocaine) performed on the facet joint medial branch block and after then RF (cobined or conventional) application under fluoroscopy.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Neuropathic Pain Scale | Scores of the patients ; before the procedure and 6 and 12 months after the procedure are shownThe 7 symptoms items are scored by interviewing the patient.The scores are added and a score of 4 or more out of ,10 point (severe pain ) .
  Neuropathic Pain 4 Questions (DN4)
Pain Rating Scale | The NRS scores of the patients before the procedure and 6 and 12 months after the procedure .NRS in which individuals rate their pain on an ten-point numerical scale. Zero:''no pain at all' ten-point ''severe pain''
  Numeric Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Nalan Celebi, Professor, Study Director — Hacettepe University; Tuğçe Yavuz, M.D, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malaithong W, Munjupong S. Combined Continuous Radiofrequency Ablation and Pulsed Neuromodulation to Treat Cervical Facet Joint Pain and Alleviate Postcervical Radiofrequency Side Effects. Anesth Pain Med. 2022 Dec 14;12(6):e129747. doi: 10.5812/aapm-129747. eCollection 2022 Dec. PMID 36938106
- [Background] Ding Y, Li H, Hong T, Zhu Y, Yao P, Zhou G. Combination of Pulsed Radiofrequency with Continuous Radiofrequency Thermocoagulation at Low Temperature Improves Efficacy and Safety in V2/V3 Primary Trigeminal Neuralgia. Pain Physician. 2018 Sep;21(5):E545-E553. PMID 30282402